CLINICAL TRIAL: NCT06093217
Title: Developing Artificial Intelligence Solutions to Improve Diagnosis and Risk Stratification in Acute Pulmonary Embolism
Brief Title: Artificial Intelligence to Improve Detection and Risk Stratification of Acute Pulmonary Embolism (AID-PE)
Acronym: AID-PE
Status: Completed | Type: Observational
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: University of Bath (Other); University of Bristol (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2720; 311735 (Other: NIHR)
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Embolism
Keywords: Artificial Intelligence; Pulmonary Embolism; CTPA; Venous Thrombo-embolic disease
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: 'Live' Introduction of AI technology: Consecutive CTPAs, for patients with suspected acute PE, which have their imaging interpreted 'live' by AI technology. The radiologist will have ultimate responsibility for the report generated.
  Interventions: Device: Artificial Intelligence
- Comparator Cohort: Standard Radiology reporting: Retrospective CTPAs, for patients with suspected acute PE, which have been reported by a human radiologist only.
  These CTPAs will not be interpreted by AI technology 'live' BUT undergo analysis to help assess the sensitivity, specificity, false negative, false positive rates of AI technology.
  Interventions: Device: Artificial Intelligence

INTERVENTIONS:
Device: Artificial Intelligence — AI technology will generate a report with relevant key slice imaging identifying the presence of an acute pulmonary embolism and RV:LV ratio measurements to the radiologist

SUMMARY:
The goal of this exploratory observational study is to assess the feasibility and real-world clinical impact of implementing Artificial Intelligence (AI) software for the detection of acute Pulmonary Embolism (PE) in patients who undergo Computed Tomography Pulmonary Angiogram (CTPA). The main questions that this study aims to answer are:

[Question 1] What is the real-world impact of AI on the clinical outcomes and decision making by radiologists and clinicians in the management of acute PE?

[Question 2] Is AI software for the detection of acute PE acceptable to use in clinical practice and do they have a favourable impact on clinical workload?

[Question 3] Is it cost-effective to implement AI software for the detection of acute PE in clinical practice?

Patients having a CTPA for the detection of acute PE will have their imaging analysed by AI software in combination with a human radiologist. Researchers will aim to compare the clinical and radiology specific outcomes with a retrospective cohort of patients who have had standard routine radiology reporting.

DETAILED DESCRIPTION:
Acute Pulmonary Embolism (PE) results from partial or total occlusion of the pulmonary blood vessels by thrombus, which can cause right ventricular failure and death if not diagnosed and treated early. Acute PE is a common condition with rising mortality. Patients with acute PE are often poorly risk stratified despite clear guidelines. In fact, the 2019 National Confidential Inquiry into Patient related Outcome and Death (NCEPOD) for acute PE highlighted the need to address worsening mortality rates through appropriate risk stratification of the condition.

ESC/ERS guidelines for the diagnosis and management of acute PE also advise on the importance of risk stratification. An increased right ventricle: left ventricle (RV:LV) ratio >1.0 on Computed Tomography Pulmonary Angiogram (CTPA) is associated 2.5-fold increased risk of all-cause mortality, and 5-fold risk for PE-related mortality. This metric is intended to help clinicians distinguish between patients with high and low risk acute PE. Patients stratified as high risk (RV:LV ratio >1.0) necessitate closer monitoring within an inpatient setting. Whereas, patients stratified as low risk (RV:LV ratio <1.0) are suitable for early discharge through ambulatory pathways.

Therefore, the provision of RV:LV metrics within radiology reporting has potentially important clinical implications. If clinicians are not provided with any quantifiable evidence of RV dysfunction on which to base their treatment decisions, patients with high risk acute PE may be unintentionally considered 'low risk' and discharged home. Furthermore, patients with low risk acute PE may be subject to longer, and potentially unnecessary, inpatient stays which undoubtedly contributes to the cost of healthcare. The integration of Artificial Intelligence (AI) technology within radiology reporting of CTPAs for acute PE could be a potential solution to address this challenge.

AI is an increasingly attractive technology within healthcare. It describes a number of computer software techniques which mimic human cognitive function. AI shows promise in ability to detect and risk stratify acute PE. However, most studies have been conducted in retrospective cohorts. Furthermore, no study current has addressed the health economic impact of implementing AI technology within the real-world reporting of acute PE.

This observational study will be led by Royal United Hospital Bath NHS Trust (RUH). The aim of this study is to integrate Artificial Intelligence and machine learning technology within the reporting of CTPAs for acute PE. The investigators hypothesise that AI technology can improve the prompt diagnosis, risk stratification, and management of acute PE within a real-world clinical setting. The investigators also hypothesis that integration of AI technology is cost-effective, and acceptable to radiologists and clinicians.

Patients whose scans will be included in the study will be all those consecutively presenting to the RUH with a possible diagnosis of acute PE for 12 months before (comparator cohort) and 12 months after (intervention cohort) 'live' introduction of integrated AI technology reporting. For all recruited participants, an anonymised clinician case report form will be used to capture details relating to their demographics, clinical-radiological PE severity, their management, and outcomes including mortality at 12 months.

At the point of analysis, the investigators will perform adjustments/matching between the two cohorts for patient baseline characteristics. The investigators will also adjust for calendar time of recruitment, to account for temporal trends. Analysis between both cohorts will also allow development of a decision analysis model to assess the cost-effectiveness of integrated AI technology within CTPA report for acute PE. Clinician and radiologist questionnaires will be used to assess user acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patient requiring CTPA to exclude or diagnose acute PE

Exclusion Criteria:

* Patients under 18 years of age
* Patients who have registered with the national opt-out scheme for research
* CTPA performed for reasons other than acute PE
* CTPA performed for acute PE but reported by external radiologists
* Incomplete or discontinued CTPA scans
* Insufficient quality CTPA to allow for analysis by a radiologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who attend the Royal United Hospital Bath NHS Trust and require CTPA to exclude or diagnose acute PE.
Sampling Method: Non-Probability Sample
Enrollment: 3872 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patient decisions made in line with evidence based best practice guidelines after introducing AI technology within CTPA reporting | 12 months
  Comparison before and after AI introduction

SECONDARY OUTCOMES:
Rate of acute PE detection with AI technology | 24 months
  True positives and True negatives
Rate of discordant acute PE cases | 24 months
  False positive and false negative rate with acute PE detection
AI failure rate for acute PE detection | 24 months
  Proportion of scans unable to be interpreted by AI despite suitable CTPA acquisition
Rate of RV:LV detection with AI technology | 24 months
  True positive and true negative
Rate of discordant RV:LV detection | 24 months
  False positive and false negative
Failure rate for automated RV:LV ratio | 24 months
  Proportion of scans unable to calculate automated RV:LV ratio despite suitable CTPA acquisition
30 day mortality | 12 months
  Patient mortality (death) at 30-days post-PE diagnosis. Comparison before and after AI introduction.
12 month mortality | 12 months
  Patient mortality (death) at 12-months post-PE diagnosis. Comparison before and after AI introduction.
Hospital admission and bed days for acute PE | 12 months
  Comparison before and after AI introduction
Time to anticoagulation in PE cases | 12 months
  Comparison before and after AI introduction
Time from CTPA to discharge | 12 months
  Comparison before and after AI introduction
PE risk stratification rates (low, intermediate low, intermediate high and high risk) | 12 months
  Comparison before and after AI introduction
Cost to NHS for acute PE | 12 months
  Comparison before and after AI introduction
End-user (clinician and radiologist) acceptability of AI technology | 12 months
  Quantified metrics from a non-validated questionnaire to evaluate end-use experience of integrated AI radiology reporting.
Referral rates to outpatient follow-up (respiratory, thrombosis, haematology) | 12 months
  Comparison before and after AI introduction
Diagnostic rate of Chronic thromboembolic pulmonary hypertension (CTEPH) | 12 months
  Comparison before and after AI introduction

OTHER OUTCOMES:
Exploratory outcomes | 12 months
  Given the exploratory nature of this observational non-randomised feasibility study, there may be patterns/outcomes which emerge/develop during the study period. The investigators will report on any patterns which may emerge following introduction of AI reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rodrigues, MBBS FRCR, Principal Investigator — Royal United Hospitals Bath NHS Foundation Trust
Locations (1):
- Royal United Hospitals, Bath NHS Foundation Trust, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided